CLINICAL TRIAL: NCT00427635
Title: A Randomized, Double-blind, Placebo Controlled, Study to Evaluate the Efficacy and Safety of Esomeprazole Once Daily for the Treatment of Gastroesophageal Reflux Disease (GERD) in Neonatal Patients, Including Premature and up to 1 Month Corrected Age
Brief Title: Efficacy and Safety of Esomeprazole Once Daily for the Treatment of GERD in Neonatal Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9614C00004
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Results first posted 2010-05-19 (Estimated); Last update posted 2010-12-20 (Estimated); Status verified 2010-12

CONDITIONS: GERD
Keywords: neonates; infants; GERD; reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole

SUMMARY:
The purpose of this study is to assess the difference between esomeprazole and placebo in the treatment of signs and symptoms as observed by 8-hour video and cardiorespiratory monitoring in neonatal patients.

ELIGIBILITY:
Inclusion Criteria:

* Full-term or gestational age >/= 28 to 44 weeks
* In-patient in Neonatal Intensive Care Unit, special care nursery, or equivalent
* Patient must be on a stable mode of feeding or with minimal variations for at least 2 days prior to randomization

Exclusion Criteria:

* Patients with a need for resectional or reconstructive surgery of the gastrointestinal tract
* Patients with any condition that may require surgery during the course of the study
* Patients with acute respiratory distress within 72 hours prior to enrollment

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2006-10; Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Illueca, MD, Study Director — AstraZeneca; Per Lundborg, MD, Study Director — AstraZeneca; Kathryn Collison, MPH, MT(ASCP), Study Director — AstraZeneca
Locations (3):
- Research Site, North Adelaide, Australia
- Research Site, Aachen, Germany
- Research Site, Sheffield, United Kingdom

REFERENCES:
- [Derived] Davidson G, Wenzl TG, Thomson M, Omari T, Barker P, Lundborg P, Illueca M. Efficacy and safety of once-daily esomeprazole for the treatment of gastroesophageal reflux disease in neonatal patients. J Pediatr. 2013 Sep;163(3):692-8.e1-2. doi: 10.1016/j.jpeds.2013.05.007. Epub 2013 Jun 22. PMID 23800403

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants either full term or those with a gestational age or post-conceptual age ³28 to 44 weeks, and who were inpatients suspected of having the following clinical findings: any 2 (either individually or in any combination) of (1) apnea +/- bradycardia +/- oxygen desaturations, (2) vomiting/gagging, (3) irritability/pain at least every second
Groups:
- Esomeprazole: Esomeprazole 0.5 mg/kg/ day once daily 30 minutes prior to a morning feeding during 15 days by oral gavage (using a nasogastric or orogastric tube) or by nippling.
- Placebo: Placebo once daily 30 minutes prior to a morning feeding during 15 days by oral gavage (using a nasogastric or orogastric tube) or by nippling.
Period: Treatment Phase
Arm/Group | Esomeprazole | Placebo
Started | 26 (Randomised) | 26 (Randomised)
Completed | 25 (ITT population. One voluntary discontinuation by parent/guardian) | 26 (ITT population)
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Study Completion to Safety Follow-up
Arm/Group | Esomeprazole | Placebo
Started | 25 | 26
Completed | 25 | 25 (One participant lost to follow-up)
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole | Placebo | Total
Number analyzed (Participants) | 26 | 26 | 52
Age Continuous [Mean (Standard Deviation); unit: Days] | 46.5 (30.3) | 46.5 (31.2) | 46.5 (30.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Normalized Number of GERD Events Observed From Video and Cardiorespiratory Monitoring
Description: The number of events are normalized prior to summary to correspond to a complete 8-hour monitoring period. Only patients with data at both baseline and final assessment are included.
Time Frame: Baseline and end of treatment (10-14 days)
Measure: Mean (Standard Deviation); unit: Mean Number of Events
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 25 | 26
Mean Number of Events | -28.01 (77.70) | -24.79 (44.25)

2. Secondary Outcome: Change From Baseline in Normalized Number of GERD Events During Video and Cardiorespiratory Monitoring Associated With Acid Reflux
Description: Event considered associated with reflux if start time of GERD sign/symptom is within 2 minutes of start time of acid reflux. The number of events are normalized prior to summary to correspond to a complete 8-hour monitoring period. Only patients with data at both baseline and final assessment are included.
Time Frame: Baseline and end of treatment (10-14 days)
Measure: Mean (Standard Deviation); unit: Mean Number of Events
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 25 | 25
Mean Number of Events | -21.79 (40.37) | -13.49 (32.76)

3. Secondary Outcome: Change From Baseline in Number of Reflux Episodes (Acid or Non-acid)
Description: Number of reflux episodes based on 24-hour impedance monitoring data
Time Frame: Baseline and end of treatment (10-14 days)
Measure: Mean (Standard Deviation); unit: Mean Number of Episodes
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 20 | 22
Mean Number of Episodes | -14.55 (49.58) | 6.27 (28.50)

4. Secondary Outcome: Change From Baseline in Number of Acidic Reflux Episodes
Description: Number of reflux episodes (pH<4.0) based on 24-hour impedance monitoring data
Time Frame: Baseline and end of treatment (10-14 days)
Measure: Mean (Standard Deviation); unit: Mean Number of Episodes
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 20 | 22
Mean Number of Episodes | -37.75 (32.38) | 2.36 (18.35)

5. Secondary Outcome: Change From Baseline in Number of Weakly Acidic Reflux Episodes
Description: Number of reflux episodes (pH 4.0-6.9) based on 24-hour impedance monitoring data
Time Frame: Baseline and end of treatment (10-14 days)
Measure: Mean (Standard Deviation); unit: Mean Number of Episodes
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 20 | 22
Mean Number of Episodes | 22.60 (45.17) | 3.59 (21.60)

6. Secondary Outcome: Change From Baseline in Number of Non Acidic Reflux Episodes
Description: Number of reflux episodes (pH>=7.0) based on 24-hour impedance monitoring data
Time Frame: Baseline and end of treatment (10-14 days)
Measure: Mean (Standard Deviation); unit: Mean Number of Episodes
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 20 | 22
Mean Number of Episodes | 0.60 (1.14) | 0.32 (0.99)

7. Secondary Outcome: Change From Baseline in Number of Liquid Acidic Reflux Episodes
Description: Number of reflux episodes based on 24-hour impedance monitoring data
Time Frame: Baseline and end of treatment (10-14 days)
Measure: Mean (Standard Deviation); unit: Mean Number of Episodes
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 20 | 22
Mean Number of Episodes | -19.00 (52.03) | 3.05 (31.19)

8. Secondary Outcome: Change From Baseline in Number of Mixed Gas/Liquid Acidic Reflux Episodes
Description: Number of reflux episodes based on 24-hour impedance monitoring data
Time Frame: Baseline and end of treatment (10-14 days)
Measure: Mean (Standard Deviation); unit: Mean Number of Episodes
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 20 | 22
Mean Number of Episodes | 4.45 (17.44) | 3.27 (13.84)

9. Secondary Outcome: Change From Baseline in Mean Bolus Clearance Time
Description: Based on 24-hour impedance monitoring data
Time Frame: Baseline and end of treatment (10-14 days)
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 20 | 22
Seconds | -0.29 (24.56) | -4.05 (25.61)

10. Secondary Outcome: Change From Baseline in Mean Acid Clearance Time
Description: Based on 24-hour impedance monitoring data
Time Frame: Baseline and end of treatment (10-14 days)
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 20 | 22
Seconds | 5.93 (64.32) | -6.36 (45.38)

11. Secondary Outcome: Change From Baseline in Percentage Time With pH<4.0
Description: Percentage time with pH<4 during 24-hour pH monitoring
Time Frame: Baseline and end of treatment (10-14 days)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 20 | 22
Percentage | -10.73 (12.63) | 2.24 (12.38)

12. Secondary Outcome: Change From Baseline in Percentage Time With pH Within 4.0-6.9
Description: Percentage time with pH 4.0-6.9 during 24-hour pH monitoring
Time Frame: Baseline and end of treatment (10-14 days)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 20 | 22
Percentage | 9.84 (12.64) | -2.60 (12.18)

ADVERSE EVENTS:
Arm/Group | Esomeprazole | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 3/7
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole (N=6) | Placebo (N=7)
Bradycardia Neonatal (Cardiac disorders) | 0 | 1
Cyanosis (Cardiac disorders) | 0 | 1
Inappropriate Device Signal Detection (Injury, poisoning and procedural complications) | 0 | 1
Infantile Apnoeic Attack (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole (N=6) | Placebo (N=7)
Anaemia Neonatal (Blood and lymphatic system disorders) | 1 | 1
Cyanosis (Cardiac disorders) | 0 | 1
Deafness Neurosensory (Ear and labyrinth disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Retinopathy Of Prematurity (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Flatulence (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Oedema Peripheral (General disorders) | 1 | 0
Neonatal Infection (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Urinary Tract Infection Neonatal (Infections and infestations) | 0 | 1
Oxygen Saturation Decreased (Infections and infestations) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less